CLINICAL TRIAL: NCT06134180
Title: An AI-Embedded Intervention to Promote Financial Wellbeing Among Latino Family Caregivers
Brief Title: CONFIDENCE-AI Financial Education for Caregivers (CONFIDENCE-AI)
Acronym: CONFIDENCE-AI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Kylie Meyer, Assistant Professor, Case Western Reserve University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY20230876
Record Dates: First submitted 2023-11-06; First posted 2023-11-18 (Actual); Results first posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Alzheimer Disease; Dementia; Caregiver Burden; Financial Stress
MeSH Terms: conditions — Alzheimer Disease; Dementia; Caregiver Burden; Financial Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CONFIDENCE AI (Experimental): Participants will attend the 4-week CONFIDENCE-AI Program. This program will include attending 4 group-based sessions delivered by videoconference. Each session will last approximately 1.5 hours each and will cover topics such as how to budget, accessing community resources to displace the out-of-pocket costs of caregiving, asking for help, and more. Participation will be supplemented by access to a digital app to support engagement, such as through text messaging and resources navigation support.
  Interventions: Behavioral: CONFIDENCE-AI

INTERVENTIONS:
Behavioral: CONFIDENCE-AI — Multicomponent psychoeducational intervention focused on financial wellbeing

SUMMARY:
The intervention being tested, CONFIDENCE-AI is a refined version of the original CONFIDENCE intervention made to reduce psychological financial strain and improve management of out-of-pocket care costs while increasing caregiver resourcefulness skills. Participants will be asked to participate in a 4-week intervention that includes participation in four, synchronous group-based Zoom sessions as well as between-session activities to apply learning. Participants will also receive tailored text message notifications from the NeuViCare AI-powered app via text and will be able to submit questions to the app to receive financial well-being information related to caregiving.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified caregiver to a person living with probable Alzheimer's disease or related dementia
* Person living with dementia meets stage 4 to 6 criteria on Global Deterioration Scale according to the family caregiver
* Has been at least 6 months since the care recipient began to experience dementia symptoms
* Latino/Hispanic ethnicity.

Exclusion Criteria:

* Individuals who plan to place their family member in a nursing home in the next 3 months
* Unreliable access to internet, tablet or smart phone, and email
* Does not agree to participate in at least 3 of the 4 group sessions and/or register for the NeuViCare app
* Unable to read and speak in English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2024-03-23 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kylie Meyer, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified survey data, such as pre- and post-test data, will be stored and available upon reasonable request with qualified investigators following the appropriate establishment of a data use agreement.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Information will be available upon study completion (i.e., once primary studies are published). De-identified data will be stored for at least 3 years following study completion.

REFERENCES:
- [Background] Zauszniewski JA, Lai CY, Tithiphontumrong S. Development and testing of the Resourcefulness Scale for Older Adults. J Nurs Meas. 2006 Spring-Summer;14(1):57-68. doi: 10.1891/jnum.14.1.57. PMID 16764178
- [Background] Ritter PL, Sheth K, Stewart AL, Gallagher-Thompson D, Lorig K. Development and Evaluation of the Eight-Item Caregiver Self-Efficacy Scale (CSES-8). Gerontologist. 2022 Mar 28;62(3):e140-e149. doi: 10.1093/geront/gnaa174. PMID 33146727
- [Background] Sadigh G, Switchenko J, Weaver KE, Elchoufi D, Meisel J, Bilen MA, Lawson D, Cella D, El-Rayes B, Carlos R. Correlates of financial toxicity in adult cancer patients and their informal caregivers. Support Care Cancer. 2022 Jan;30(1):217-225. doi: 10.1007/s00520-021-06424-1. Epub 2021 Jul 13. PMID 34255179

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CONFIDENCE AI
Started | 14
Completed Baseline | 14
Completed First Follow up Survey | 11
Completed Second Follow up Survey | 10
Completed | 10 (14 caregivers enrolled and completed the baseline survey. 11 complted the first follow up survey. 10 completed the second follow up survey.)
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | CONFIDENCE AI
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 2
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 14
Financial Strain [Mean (Standard Deviation); unit: units on a scale] — Population: One participant skipped a survey item at baseline required to calculate financial strain score.
  units on a scale
    number analyzed (Participants) | 13
    (all) | 28.4 (5.6)
Resourcefulness [Mean (Standard Deviation); unit: units on a scale] — Population: One caregiver skipped a survey item required to calculate a score on this measure at baseline.
  units on a scale
    number analyzed (Participants) | 13
    (all) | 75.3 (34.1)
Self-Efficacy [Mean (Standard Deviation); unit: units on a scale] | 32.0 (16.7)

OUTCOME MEASURES:

1. Primary Outcome: Financial Strain
Description: Financial strain will be measured using the 11-item Comprehensive Score for Financial Toxicity (COST) Scale. A modified version of COST demonstrates validity and reliability when tested among cancer caregivers (α=0.91; range: 0 to 44). COST items are generic enough to be applicable to caregivers to persons PLWD without further modification (e.g., "I feel financially stressed"). Caregivers are asked to indicate if each statement applies to them "Not at all" (0) to "Very much" (4). Higher scores indicate higher levels of financial strain.
Time Frame: The outcome measure will use the average change score from baseline scores until post-intervention (1 month post-baseline) and 2 months post-intervention (3-months after the baseline).
Population: From baseline to the post-intervention data collection point, three participants were lost to follow up and one participant was missing a survey item response required to calculate this score. Thus, data is available for 10 of 14 participants.
  From baseline to the 2-month post-intervention data collection point, one more case was lost to follow up and another was missing a survey item response required to calculate this score. Thus, data is available for 9 of 14 participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CONFIDENCE AI
Number analyzed (Participants) | 10
units on a scale
  Change score from baseline scores until post-intervention | -3.4 (4.9)
  Change score from baseline scores until 2-months post-intervention: number analyzed (Participants) | 9
  Change score from baseline scores until 2-months post-intervention | -4.7 (6.6)

2. Primary Outcome: Resourcefulness
Description: Resourcefulness is measured using the 28-item Caregiver Resourcefulness Scale (alpha=0.85). This scale has two factors: one focused on help-seeking and another on self-help. Caregivers are asked the frequency at which they use different strategies to manage challenges, and may respond: Not at all like me (0), Pretty much not like me (1), A little bit not like me (2), A little bit like me (3), Pretty much like much like me (4), or Very much like me (5). Items are added together to create a total score. Scores range from 0 to 140, where higher scores indicate higher levels of resourcefulness. The outcome measure will use the average change score from baseline scores
Time Frame: as for outcome 1
Population: From baseline to the post-intervention data collection point, three participants were lost to follow up and one participant was missing a survey item response required to calculate this score. Thus, data is available for 10 of 14 participants.
  From baseline to the 2-month post-intervention data collection point, one more case was lost to follow up and two more cases were missing a survey item response required to calculate this score. Thus, data is available for 8 of 14 participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CONFIDENCE AI
Number analyzed (Participants) | 14
score on a scale
  Change score from baseline scores until post-intervention: number analyzed (Participants) | 10
  Change score from baseline scores until post-intervention | 13.2 (25.7)
  Change score from baseline scores until 2-months post-intervention: number analyzed (Participants) | 8
  Change score from baseline scores until 2-months post-intervention | 11.3 (13.3)

3. Secondary Outcome: Self-Efficacy
Description: Self-efficacy is measured using the Caregiver Self-Efficacy Scale. This 8-item scale asks about multiple domains of self-efficacy (e.g., managing behavioral symptoms, accessing respite, and controlling upsetting thoughts). It demonstrates high reliability (alpha=0.89) and good test-retest reliability (0.73). Participants rate the extent to which they are "Not confident at all" (1) to "Totally confident" (10). Scores range from 8 (lowest level of self-efficacy) to 80 (highest level of self-efficacy).
Time Frame: as for outcome 1
Population: From baseline to the post-intervention data collection point, three participants were lost to follow up. Thus, data is available for 10 of 14 participants.
  From baseline to the 2-month post-intervention data collection point, one more case was lost to follow up and another was missing a survey item response required to calculate this score. Thus, data is available for 9 of 14 participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CONFIDENCE AI
Number analyzed (Participants) | 14
units on a scale
  Change score from baseline scores until post-intervention: number analyzed (Participants) | 11
  Change score from baseline scores until post-intervention | 16.3 (15.2)
  Change score from baseline scores until 2-months post-intervention: number analyzed (Participants) | 9
  Change score from baseline scores until 2-months post-intervention | 13.2 (10.3)

ADVERSE EVENTS:
Time Frame: Through study completion, approximately 4 months
Groups:
- CONFIDENCE-AI: Participants will attend the 4-week CONFIDENCE-AI Program. This program will include attending 4 group-based sessions delivered by videoconference. Each session will last approximately 1.5 hours each and will cover topics such as how to budget, accessing community resources to displace the out-of-pocket costs of caregiving, asking for help, and more. Participation will be supplemented by access to a digital app to support engagement, such as through text messaging and resources navigation support.
Arm/Group | CONFIDENCE-AI
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-19): https://cdn.clinicaltrials.gov/large-docs/80/NCT06134180/Prot_SAP_000.pdf
  • Informed Consent Form (2024-11-03): https://cdn.clinicaltrials.gov/large-docs/80/NCT06134180/ICF_001.pdf